CLINICAL TRIAL: NCT00004141
Title: Phase II Study of Outpatient CDDP and DTIC Followed by GM-CSF, IFN-a2b, and IL-2 in Patients With Advanced Melanoma
Brief Title: Combination Chemotherapy Plus Biological Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9372; UCCRC-9372; UCCRC-CTRC-9821; NCI-G99-1615
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Cisplatin; Dacarbazine; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): CDDP (75 mg/m2) and DTIC (660 mg/m2) will be administered sequentially by intravenous infusion in day 1. Subsequently, GM-CSF (450 mg/ m2) will be administered SC days 2-7; IL-2 (11 MU daily) will be given SC days 8-14, and IFN-2b (9 MU) will be given SC days 8, 10, 12, and 14.
  Interventions: Drug: Cisplatin; Drug: dacarbazine; Drug: Granulocyte-macrophage colony-stimulating factor

INTERVENTIONS:
Drug: Cisplatin
  Other Names: CDDP
Drug: dacarbazine
  Other Names: DTIC
Drug: Granulocyte-macrophage colony-stimulating factor
  Other Names: GM-CSF

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies use different ways to stimulate the immune system and stop cancer cell from growing. Combining more than one drug with different types of biological therapies may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus biological therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of cisplatin and dacarbazine followed by sargramostim (GM-CSF), interferon alfa, and interleukin-2 in patients with metastatic melanoma.
* Determine the objective response rate, relapse free survival, and overall survival of these patients on this regimen.

OUTLINE: Patients receive cisplatin IV over 1 hour and dacarbazine IV over 30-60 minutes sequentially on day 1, followed by sargramostim (GM-CSF) subcutaneously (SC) on days 2-7, interleukin-2 SC on days 8-14, and interferon alfa SC on days 8, 10, 12, and 14. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression, and then every 8-12 weeks thereafter.

PROJECTED ACCRUAL: A total of 15-45 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma

  * Stage III with intransit metastases
  * Stage IV
* No uncontrolled brain metastases by CT scan
* No clinically significant ascites or pleural effusions

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 10 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.5 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT no greater than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 70 mL/min

Cardiovascular:

* No clinically significant cardiac disease on EKG, echocardiogram, or MUGA scan

Pulmonary:

* No clinically significant pulmonary disease on chest x-ray

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant thyroid dysfunction
* No concurrent severe infection
* No other medical or psychiatric condition that would interfere with compliance
* No second malignancy within the past 5 years, except:

  * Localized nonmelanomatous skin cancer
  * Carcinoma in situ of the cervix
  * Grade 1 Ta bladder cancer
* Suspected hearing deficits must undergo audiologic testing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than one prior immunotherapy regimen
* At least 4 weeks since prior immunotherapy
* Adjuvant interferon alfa before relapse allowed

Chemotherapy:

* No more than one prior chemotherapy regimen
* At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas)
* No concurrent cyclophosphamide
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroids or cyclosporine A

Radiotherapy:

* At least 2 weeks since prior radiotherapy

Surgery:

* At least 3 weeks since major surgery

Other:

* No concurrent immunosuppressive drugs
* No other concurrent investigational antineoplastic drugs
* Concurrent thyroid replacement therapy allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1998-08; Primary Completion 2003-01 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Gajewski, MD, PhD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States